CLINICAL TRIAL: NCT04464876
Title: SATURN Transcatheter Mitral Valve Replacement for Functional Mitral Regurgitation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: InnovHeart (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TP-0050
Record Dates: First submitted 2020-06-24; First posted 2020-07-09 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-01

CONDITIONS: Mitral Regurgitation; Valve Heart Disease; Heart Valve Diseases; Mitral Valve Disease; Mitral Disease
MeSH Terms: conditions — Mitral Valve Insufficiency; Heart Valve Diseases; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): SATURN TA TMVR Device implanted
  Interventions: Device: SATURN TA System

INTERVENTIONS:
Device: SATURN TA System — SATURN TA TMVR Device implanted

SUMMARY:
This study is a prospective, single-arm, multi-center feasibility clinical study of the SATURN TA System for the treatment of NYHA Class ≥ II patients with severe functional mitral regurgitation who are not suitable for surgical treatment following Heart Team assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older.
2. Severe functional mitral regurgitation (≥ Grade 3+).
3. NYHA functional Class ≥ II. If Class IV, patient must be ambulatory.
4. Treatment and compliance with optimal guideline-directed medical therapy (GDMT) for heart failure for at least 30 days.
5. Not a suitable candidate for open mitral valve surgery due to high operative risk, as determined by the Heart Team.
6. Able to complete quality-of-life assessment (KCCQ).

General Exclusion Criteria:

1. Excessive frailty or comorbid conditions that preclude the anticipated benefit of the valve replacement.
2. Life expectancy <1 yr due to noncardiac conditions.
3. Active endocarditis.
4. Active systemic infection.
5. Modified Rankin Scale ≥4 disability.
6. Hemodialysis/ chronic renal failure (eGFR < 35 mL/min/m2).
7. Pulmonary arterial hypertension (fixed PAS < 60mmHg). 8) COPD on home oxygen.

9) Refuses blood transfusions. 10) Documented bleeding or coagulation conditions (hypo- or hyper-coagulable states).

11) Severe connective tissue disease under chronic immunosuppressive or cortisone therapy.

12) Pregnant/ lactating. Females of childbearing age must be willing to take contraceptives.

13) Participating in other investigational studies likely to confound the results or affect the study.

14) Unable to consent. 15) Unable or unwilling to comply with study Follow-up. 16) Patients classified as "vulnerable patients".

Cardiovascular Exclusion Criteria:

1. Myocardial infarction during prior 30 days.
2. Stroke or TIA during prior 30 days.
3. Severe extracardiac arteriopathy (safety measure for extra-circulatory support if surgical conversion is needed).
4. Prior mitral valve treatment (e.g. valve repair or replacement, MitraClip, etc.), and/or anticipated mitral valve treatment prior to enrollment.
5. Prior surgical mechanical valve AVR.
6. Prior TAVI.
7. Need for any cardiovascular surgery or intervention (other than for MV disease) within 30 days.
8. CRT or ICD implanted in previous 30 days.
9. Cardiogenic shock, hemodynamic instability, Systolic Blood Pressure <90mmHg, Inotropic dependent or IABP/mechanical circulatory support.
10. CABG or PCI within previous 30 days.
11. Adequately treated for cardiac condition per applicable standards, such as for coronary artery disease, left ventricular dysfunction, mitral regurgitation, or heart failure. No need for revascularization.
12. Prior or planned heart transplantation (UNOS status 1).
13. Physical evidence of right-sided congestive heart failure:

    1. Patients with ascites.
    2. Patients with anasarca (generalized edema / hydropsy).

    Procedural Exclusion Criteria:
14. Chest condition that prevents transapical access.
15. Known hypersensitivity or contraindication to procedural or post-procedural medication (e.g., contrast solution, anticoagulation therapy).
16. Documented hypersensitivity to nickel or titanium.

Cardiac Exclusion Criteria (evaluated by Core Labs):

1. Left ventricular EF ≤ 30% by imaging.
2. Severe mitral annular calcification, severe mitral stenosis, valvular vegetation or mass.
3. Extensive mitral flail leaflets.
4. Left ventricular thrombus, mass, or vegetation.
5. Left ventricular end-diastolic diameter > 7.5 cm.
6. Severe right ventricular dysfunction.
7. Significant intracardiac shunt.
8. Anatomic ineligibility for SATURN valve as determined by the Screening Committee.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-08-19 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Freedom from device-related or procedure-related major adverse events | 30 days
  Freedom from device-related or procedure-related major adverse events at 30 days (cardiac death, peri-procedural myocardial infarction, disabling stroke, renal failure requiring dialysis, life threatening bleeding).
Reduction of mitral regurgitation | 30 days
  Reduction of mitral regurgitation to ≤1 at 30 days.
Technical success | Day 0
  Technical success defined as alive patient at exit from procedure room, with all of the following:
  * Successful access, delivery and retrieval of the delivery systems.
  * Development and correct positioning of the bioprosthesis.
  * Freedom of additional emergency surgery or re-intervention related to the device or access procedure.

SECONDARY OUTCOMES:
Freedom from device-related or procedure-related major adverse events | 30 days, 1 year, 2 years
  * Freedom from device-related or procedure-related major adverse events throughout long- term follow-up.
  * Freedom from all-cause mortality
Freedom from all-cause mortality | 30 days, 1 year, 2 years
  Freedom from all-cause mortality
Patients success | 30 days, 1 year, 2 years
  Patients success
Device success | 30 days, 1 year, 2 years
  Device success
6 Minute Hall Walk Test | 30 days, 1 year, 2 years
  Improvement from baseline in functional status by ≥ 30 meters
KCCQ | 30 days, 1 year, 2 years
  Improvement from baseline in Quality of Life by ≥ 10 points.
NYHA functional classification | 30 days, 1 year, 2 years
  Improvement from baseline by ≥ 1 functional classification.

CONTACTS AND LOCATIONS:
Overall Officials: Marie Steinbrink, Study Director — InnovHeart
Locations (3):
- Rigshospitalet University Hospital of Copenhagen, Copenhagen, Denmark
- Heart And Vascular Center, Semmelweis University, Budapest, Hungary
- Vilnius University Hospital Santaros klinikos, Vilnius, Lithuania

IPD SHARING:
Plan to Share IPD: No